CLINICAL TRIAL: NCT00977223
Title: Pilot Study of the Action of the Substance P Antagonist Aprepitant on Aldosterone and Cortisol Secretion in Healthy Volunteers.
Brief Title: Effects of Substance P Antagonists on Adrenal Secretion
Acronym: APHOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 2007/049/HP; 2008-003367-40 (EudraCT Number)
Record Dates: First submitted 2009-09-14; First posted 2009-09-15 (Estimated); Last update posted 2012-02-16 (Estimated); Status verified 2012-02

CONDITIONS: Healthy Volunteers
Keywords: Aldosterone; Substance P; Cortisol; Aprepitant; Adrenal glands
MeSH Terms: interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aprepitant (Experimental): 7 days treatment with study drug, order of periods (active treatment or placebo) being sorted out.
  Interventions: Drug: aprepitant/placebo
- placebo (Placebo Comparator): 7 days treatment with study drug, order of periods (active treatment or placebo) being sorted out.
  Interventions: Drug: aprepitant/placebo

INTERVENTIONS:
Drug: aprepitant/placebo — Aprepitant, 125 MG at day 1 then 80 MG day 2-7, once a day, per os, at 8 AM during breakfast
  Other Names: DCI : Aprepitant; Brand name : Emend

SUMMARY:
Data from the literature and previous in vitro research conducted in the investigators' laboratory (INSERM U413/EA4310, University of Rouen) suggest that adrenal corticosteroid secretion might be controlled by sympathetic nervous system. This neurocrine regulation of corticosteroid secretion involves locally released neuropeptides. Among them, substance P is able to stimulate aldosterone and cortisol production via NK1 receptors.

The aim of the present study is to investigate the effects of a NK1 receptor antagonist, aprepitant, on adrenocortical secretions in healthy volunteers. Aprepitant is a drug already available for the treatment of nausea induced by chemotherapy.

In the present phase IV trial, plasma aldosterone and cortisol levels will be measured under treatment with aprepitant versus placebo, in both basal conditions and after activation of the adrenocortical function by various stimuli, including upright posture, metoclopramide, and insulin-induced hypoglycaemia. All healthy volunteers will be given the two substances (aprepitant and placebo) in a random order during two one-week periods separated by a 14 day-wash-out.

This study should allow to determine the role of substance P in the control of corticosteroid production in normal man.

DETAILED DESCRIPTION:
STUDY DESIGN

Phase IV, proof of concept, interventional, monocentric, randomised, double blind, cross-over study: The effects of a substance P antagonist (Emend) on corticosteroid secretion will be compared to those of a placebo.

STUDY OBJECTIVES

Main objective: to verify that adrenal corticosteroid secretion is actually controlled by substance P.

Secondary objective: to determine the physiological conditions that involve the control of adrenocortical function by tachykinins.

NUMBER OF SUBJECTS

20 healthy volunteers

ELIGIBILITY CRITERIA

(see below)

DURATION OF STUDY

Overall duration: 13 months Inclusion period: 12 months Follow up period (for 1 subject): 5 weeks Exclusion period: 1 month

ENDPOINTS

PRIMARY ENDPOINT: blood aldosterone variation during orthostatic test

SECONDARY ENDPOINTS

Basal aldosterone alteration Aldosterone variation during metoclopramide & hypoglycaemia tests Basal and stimulated (3 different tests) alterations of renin, cortisol & ACTH

REGULATORY AUTHORIZATIONS

Ethics committee authorization: dec 18th, 2008 Regulatory authorization: march 3rd, 2009

ELIGIBILITY:
Inclusion Criteria:

* Male subjects;
* Age ranging 18 - 30 years old;
* Submitted to a social security regimen;
* Agreeing to the study & Informed consent form signed;
* Body mass index ([weight (kg)/height (m)]²) < 27;
* No treatment received 6 weeks before inclusion;
* No anomaly after: complete clinical examination, pulse and blood pressure measurement, ECG;
* No biological abnormality after the following biological testing:

  * Hematology: white & red blood cells & platelets count, haemoglobin, hematocrit
  * Blood biochemistry: sodium, potassium, chloride, bicarbonate, creatinine, urea
  * Urinary biochemistry (24 h collection): cortisol, aldosterone
  * Serologies: HIV, HBV, HCV
* No participation in a clinical trial 3 months before inclusion.

Exclusion Criteria:

* Subject not agreeing to the study or impossible to follow-up;
* Known history of significant medical or surgical pathology, notably endocrine;
* Renal or hepatic insufficiency;
* Nephrotic syndrome;
* Edematous syndrome;
* Hypertension or postural hypotension;
* Cardiac rhythm or conduction pathologies;
* Cardiac insufficiency;
* Epilepsy;
* Significant psychiatric disorder;
* Known history of severe allergy, hypersensitivity to aprepitant ant/or metoclopramide;
* Hereditary problems of fructose intolerance, glucose-galactose malabsorption or sucrase-isomaltase deficit;
* Impaired lactose tolerance.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-06; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Plasma aldosterone variation during orthostatic test | Day 5 of treatment, at each period

SECONDARY OUTCOMES:
Basal aldosterone alteration; Aldosterone variation during metoclopramide & hypoglycaemia tests; Basal and stimulated (3 different tests) alterations of renin, cortisol & ACTH | Day 4, 5 and 7 of treatment, at each period

CONTACTS AND LOCATIONS:
Overall Officials: Hervé Lefebvre, PHD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen Clinical research Centre (CIC 0204), Rouen, Haute Normandie, France

REFERENCES:
- [Derived] Wils J, Duparc C, Cailleux AF, Lopez AG, Guiheneuf C, Boutelet I, Boyer HG, Dubessy C, Cherifi S, Cauliez B, Gobet F, Defortescu G, Menard JF, Louiset E, Lefebvre H. The neuropeptide substance P regulates aldosterone secretion in human adrenals. Nat Commun. 2020 May 29;11(1):2673. doi: 10.1038/s41467-020-16470-8. PMID 32471973